CLINICAL TRIAL: NCT02300103
Title: An Open Label Study to Evaluate The Efficacy And Safety Of Sofosbuvir/GS-5816 Fixed Dose Combination With Ribavirin For 24 Weeks In Chronic HCV Infected Subjects Who Participated In A Prior Gilead Sponsored HCV Treatment Study
Brief Title: Efficacy And Safety Of Sofosbuvir/Velpatasvir Fixed Dose Combination With Ribavirin in Chronic HCV Infected Adults Who Participated in a Prior Gilead Sponsored HCV Treatment Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-342-1553
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Results first posted 2017-07-28 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2017-06

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SOF/VEL+RBV (Experimental): Participants will receive SOF/VEL fixed dose combination (FDC) and RBV for 24 weeks.
  Interventions: Drug: SOF/VEL; Drug: RBV

INTERVENTIONS:
Drug: SOF/VEL — 400/100 mg FDC tablet administered orally once daily
  Other Names: GS-7977/GS-5816; Epclusa®
Drug: RBV — Tablet (s) administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)

SUMMARY:
The primary objective of this study is to evaluate the efficacy, safety and tolerability of treatment with sofosbuvir/velpatasvir (Epclusa®; SOF/VEL) with ribavirin (RBV) for 24 weeks in adults with chronic hepatitis C virus (HCV) infection who participated in a prior Gilead sponsored study and did not achieve sustained virologic response (SVR).

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to provide written informed consent
* HCV genotype determined by the Central Laboratory
* HCV RNA > LLOQ at screening
* Participated and completed a Gilead sponsored HCV treatment study of direct acting antiviral (DAA) containing regimens.
* Male and female of childbearing potential must agree to use protocol specified method(s) of contraception

Key Exclusion Criteria:

* Current or prior history: Clinically-significant illness (other than HCV) or any other major medical disorder that may interfere with treatment, assessment or compliance with the protocol; individuals currently under evaluation for a potentially clinically-significant illness (other than HCV) are also excluded.
* Screening ECG with clinically significant abnormalities
* Laboratory results outside of acceptable ranges at screening
* Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2016-07-02 (Actual); Study Completion 2016-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (30):
- United States (23):
  - San Diego, California
  - San Marcos, California
  - Aurora, Colorado
  - Gainesville, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Wellington, Florida
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Hillsborough, New Jersey
  - Manhasset, New York
  - Durham, North Carolina
  - Fayetteville, North Carolina
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - San Antonio, Texas
  - Falls Church, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
- Australia (4):
  - Darlinghurst, New South Wales
  - Fitzroy, Victoria
  - Melbourne, Victoria
  - Murdoch, Western Australia
- New Zealand (2):
  - Auckland
  - Christchurch
- San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Result] Gane EJ, Shiffman ML, Etzkorn K, Morelli G, Stedman C, Davis MN, et al. Sofosbuvir/Velpatasvir in Combination With Ribavirin for 24 Weeks is Effective Retreatment for Patients Who Failed Prior NS5A Containing DAA Regimens: Results of the GS-US-342-1553 Study [Abstract PS024]. J Hepatology 2016;64:S147-S8.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 31 study sites in North America and Asia Pacific. The first participant was screened on 01 December 2014. The last study visit occurred on 15 September 2016.
Pre-assignment Details: 74 participants were screened.
Groups:
- SOF/VEL+RBV: Sofosbuvir/velpatasvir (Epclusa®; SOF/VEL) (400/100mg) fixed-dose combination (FDC) tablet once daily + ribavirin (RBV) tablets (1000 mg or 1200 mg) for 24 weeks
Period: Overall Study
Arm/Group | SOF/VEL+RBV
Started | 69
Completed | 63
Not Completed | 6
Not completed — Lack of Efficacy | 3
Not completed — Protocol Violation | 1
Not completed — Withdrew Consent | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who received at least 1 dose of study drug
Groups:
- SOF/VEL+RBV: SOF/VEL (400/100mg) FDC tablet once daily + RBV tablets (1000 mg or 1200 mg) for 24 weeks
Arm/Group | SOF/VEL+RBV
Number analyzed (Participants) | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 53
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 3
  White | 61
  Asian | 2
  Native Hawaiian or Pacific Islander | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 64
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35
  New Zealand | 29
  Australia | 5
IL28b Status [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 23
    CT | 32
    TT | 14
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.4 (0.67)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 15
  ≥ 800,000 IU/mL | 54

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 is defined as HCV RNA < the lower limit of quantitation (LLOQ) 12 weeks following the last dose of study drug.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: all enrolled participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL+RBV
Number analyzed (Participants) | 69
percentage of participants | 91.3 [82.0 to 96.7]

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to 24 weeks
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL+RBV
Number analyzed (Participants) | 69
percentage of participants | 5.8

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR24 are defined as HCV RNA < LLOQ at 4 and 24 weeks following the last dose of study drug.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL+RBV
Number analyzed (Participants) | 69
percentage of participants
  SVR4 | 92.8 [83.9 to 97.6]
  SVR24 | 89.9 [80.2 to 95.8]

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ On-treatment
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL+RBV
Number analyzed (Participants) | 69
percentage of participants
  Week 1 | 15.9 [8.2 to 26.7]
  Week 2 | 60.9 [48.4 to 72.4]
  Week 4 | 91.3 [82.0 to 96.7]
  Week 6: number analyzed (Participants) | 68
  Week 6 | 98.5 [92.1 to 100.0]
  Week 8: number analyzed (Participants) | 68
  Week 8 | 97.1 [89.8 to 99.6]
  Week 12: number analyzed (Participants) | 67
  Week 12 | 98.5 [92.0 to 100.0]
  Week 16: number analyzed (Participants) | 66
  Week 16 | 100.0 [94.6 to 100.0]
  Week 20: number analyzed (Participants) | 66
  Week 20 | 100.0 [94.6 to 100.0]
  Week 24: number analyzed (Participants) | 66
  Week 24 | 100.0 [94.6 to 100.0]

5. Secondary Outcome: HCV RNA Change From Baseline
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL+RBV
Number analyzed (Participants) | 69
log10 IU/mL
  Week 1: number analyzed (Participants) | 68
  Week 1 | -4.45 (0.615)
  Week 2: number analyzed (Participants) | 67
  Week 2 | -5.04 (0.685)
  Week 4: number analyzed (Participants) | 68
  Week 4 | -5.18 (0.719)
  Week 6: number analyzed (Participants) | 68
  Week 6 | -5.23 (0.669)
  Week 8: number analyzed (Participants) | 67
  Week 8 | -5.23 (0.675)
  Week 12: number analyzed (Participants) | 66
  Week 12 | -5.23 (0.679)
  Week 16: number analyzed (Participants) | 66
  Week 16 | -5.23 (0.679)
  Week 20: number analyzed (Participants) | 66
  Week 20 | -5.23 (0.679)
  Week 24: number analyzed (Participants) | 66
  Week 24 | -5.23 (0.679)

6. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as:
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL+RBV
Number analyzed (Participants) | 69
percentage of participants | 7.2

ADVERSE EVENTS:
Time Frame: Treatment Phase: Up to 24 weeks with an onset date on or after the study drug start date plus 30 days
Description: Safety Analysis Set
Arm/Group | SOF/VEL+RBV
All-Cause Mortality (participants affected / at risk) | 0/69
Serious Adverse Events (participants affected / at risk) | 1/69
Other Adverse Events (participants affected / at risk) | 55/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL+RBV (N=69)
Nephrolithiasis (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL+RBV (N=69)
Haemolytic anaemia (Blood and lymphatic system disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 15
Vomiting (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 22
Upper respiratory tract infection (Infections and infestations) | 9
Viral upper respiratory tract infection (Infections and infestations) | 6
Headache (Nervous system disorders) | 12
Insomnia (Psychiatric disorders) | 11
Irritability (Psychiatric disorders) | 9
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 10
Rash (Skin and subcutaneous tissue disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years